CLINICAL TRIAL: NCT00921232
Title: Crossed Assessment of the Burden Within the Dyad Patient/Caregiver: Analysis of Explanatory Factors and Consequences for Return at Home of the Life-ending Patient
Brief Title: Assessment of the Burden Within the Dyad Patient/Caregiver
Acronym: RAPSODIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Unité de REcherche en sciences Cognitives et Affectives URECA EA1059 (Unknown); University of Lille Nord de France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RAPSODIE; NCT00958594 (obsolete NCT alias)
Record Dates: First submitted 2009-05-29; First posted 2009-06-16 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Palliative Care
Keywords: Life-ending patient; caregiver
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dyad (Other): life-ending patient and its caregiver
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — During a consultation:
  * 3 questionnaires (HADS, FRI, CRA)
  * and a form for the sociodemographic data

SUMMARY:
This study is about the patients life ending and their caregiver, when a return to home is planned.

This is a behavioral sciences study (= interventional study for french law)

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Cancer for which no curative treatment is envisaged
* Palliative treatment only
* For the caregiver: designated by the patient like the referring individual

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Caregiver Reaction Assessment (CRA scale) completed by patient (hetero-perception) and its caregiver (auto-perception) | At baseline, to the announcement of the exclusive palliative care

SECONDARY OUTCOMES:
Perception of the burden by the patient and its caregiver: search for potential predictive factors of the burden by statistic analysis HADS (The Hospital Anxiety and Depression Scale FRI (The Family Relationship Index) | At baseline, to the announcement of the exclusive palliative care
Search for factors influencing the return at home of the life-ending patients by statistic analysis | Death

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France